CLINICAL TRIAL: NCT01071902
Title: Safety and Efficacy Evaluation of Topical Moxidex Otic Solution in the Treatment of Acute Otitis Media With Otorrhea in Tympanostomy Tubes
Brief Title: Safety and Efficacy of Moxidex Otic
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Management decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-09-033
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Acute Otitis Media
Keywords: ear tubes; ear drainage; ear infection; ear drops; acute otitis media
MeSH Terms: conditions — Otitis Media; Otitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Moxidex (Experimental): Moxidex otic solution
  Interventions: Drug: Moxidex otic solution; Device: Tympanostomy tubes
- Moxifloxacin (Active Comparator): Moxifloxacin otic solution
  Interventions: Drug: Moxifloxacin otic solution; Device: Tympanostomy tubes
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Other: Vehicle; Device: Tympanostomy tubes

INTERVENTIONS:
Drug: Moxidex otic solution — 4 drops into the infected ear(s) twice daily (morning and evening) for 7 days
  Arms: Moxidex
Drug: Moxifloxacin otic solution — 4 drops into the infected ear(s) twice daily (morning and evening) for 7 days
  Arms: Moxifloxacin
Other: Vehicle — 4 drops into the infected ear(s) twice daily (morning and evening) for 7 days
  Arms: Vehicle
Device: Tympanostomy tubes — Tubes surgically inserted through the ear drum for the treatment of recurrent otitis media in children

SUMMARY:
The purpose of this study is to determine if Moxidex otic solution is safe and effective in treating middle ear infections in patients with ear tubes.

ELIGIBILITY:
Inclusion Criteria:

* 6 months to 12 years of age
* Ear tubes in one or both ears
* Ear drainage visible by parent/guardian
* Ear drainage less than 21 days
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Patients not otorrhea-free for 7 or less following tympanostomy tube surgery
* Ear tube with antimicrobial activity; ear tube longer than 2.5mm
* Non-tube otorrhea
* No otic surgery other than tube placement in the last year
* No menarchial females; no diabetic patients
* No patients with any disease or condition that would negatively affect the conduct of the study
* No patients taking any other systemic antimicrobial therapy during the study
* Patient must meet certain medication washouts to be eligible
* Analgesic use (other than acetaminophen) is not allowed
* Patients may not be predisposed to neurosensory hearing loss
* Other protocol-defined exclusion criteria may apply

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Clinical Cure at End of Treatment | Day 8

SECONDARY OUTCOMES:
Time to Cessation of Otorrhea | From First Dose
Microbiological Success at End of Treatment | Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Contact Alcon Call Center, Study Director — 1-888-451-3937
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States